CLINICAL TRIAL: NCT01242033
Title: An Acute Intervention Study Investigating the Effect of Red Raspberry Consumption on Post-prandial Oxidative Stress
Brief Title: Effect of Acute Red Raspberry Consumption on Post-prandial Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Dr AV Rao, PhD, Professor Emeritus, Department of Nutritional Sciences, Faculty of Medicine, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 24774
Record Dates: First submitted 2010-11-08; First posted 2010-11-16 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-11

CONDITIONS: Oxidative Stress; Antioxidants
Keywords: red raspberries; post-prandial; oxidative stress; antioxidants; polyphenols; vitamin C; acute dietary intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- one cup red raspberries (Experimental): treatment meal consists of one cup red raspberries
  Interventions: Dietary Supplement: red raspberries
- two cups red raspberries (Experimental): treatment meal consists of two cups red raspberries
  Interventions: Dietary Supplement: red raspberries
- four cups red raspberries (Experimental): treatment meal consists of four cups red raspberries
  Interventions: Dietary Supplement: red raspberries
- bread (Placebo Comparator): treatment meal consists of two slices white bread
  Interventions: Dietary Supplement: bread controls
- vitamin C (Active Comparator): treatment meal consists of two slices white bread and 200 mg vitamin C in the form of supplemental ascorbic acid
  Interventions: Dietary Supplement: bread controls

INTERVENTIONS:
Dietary Supplement: red raspberries — single serving of one, two or four cups red raspberries
  Arms: four cups red raspberries; one cup red raspberries; two cups red raspberries
Dietary Supplement: bread controls — two slices white bread alone or with 200 mg vitamin C supplement
  Arms: bread; vitamin C

SUMMARY:
Eight healthy adult subjects will be given a meal of one, two or four cups red raspberries, or two slices white bread with or without 200 mg vitamin C, after an overnight fast and consumption of a low polyphenol diet for two days. Blood samples will be taken at various time points over an eight hour period to measure oxidative stress and antioxidant levels in the blood. Each subject will attend 5 study visits with one week intervals and be given each meal in a random order. It is hypothesized that raspberry consumption at higher doses will greater protect against meal-induced oxidative stress compared to bread controls.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* blood pressure greater than 120/80 mm Hg
* body mass index greater than 24.9 kg/m^2
* history of any chronic disease
* currently taking medications
* allergy to fruit

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
change in antioxidant capacity from baseline (-0.25 h) | -0.25, 0.25, 0.5, 1, 2, 4 hours post-intake
  plasma antioxidant capacity measured using the 2,2'-azino-bis(3-ethylbenzthiazoline-6-sulphonic acid) (ABTS) radical cation assay and expressed in Trolox Equivalents (TE)

SECONDARY OUTCOMES:
change in lipid peroxidation from baseline (-0.25 h) | -0.25, 0.25, 0.5, 1, 2, 4 hours post-intake
  serum thiobarbituric acid reactive substances (TBARS) measured as an indicator of the lipid peroxidation product malondialdehyde (MDA)
change in thiols compared to baseline (-0.25 h) | -025, 0.25, 0.5, 1, 2, 4 hours post-intake
  plasma thiols quantified by 5,5'-dithiobis-(2-nitrobenzoic acid) (DTNB) assay as an indicator of the level of protection against protein oxidation

CONTACTS AND LOCATIONS:
Overall Officials: A V Rao, PhD, Principal Investigator — University of Toronto
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre; St. Michael's Hospital, Toronto, Ontario, Canada